CLINICAL TRIAL: NCT00099801
Title: Safety and Efficacy of FTY720 in Adult Patients Who Receive a Kidney Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720A2307
Record Dates: First submitted 2004-12-21; First posted 2004-12-21 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Kidney Transplantation
Keywords: Kidney, Transplantation, Rejection, Immunosuppression
MeSH Terms: conditions — Rejection, Psychology | interventions — Fingolimod Hydrochloride

INTERVENTIONS:
Drug: FTY720

SUMMARY:
The safety and efficacy of FTY720 is being evaluated in patients who receive a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing their first kidney transplant
* Male or female age 18 to 65 years

Exclusion Criteria:

* Patients in need of second kidney transplant or multi-organ transplants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis

REFERENCES:
- [Result] Saab G, Almony A, Blinder KJ, Schuessler R, Brennan DC. Reversible cystoid macular edema secondary to fingolimod in a renal transplant recipient. Arch Ophthalmol. 2008 Jan;126(1):140-1. doi: 10.1001/archophthalmol.2007.23. No abstract available. PMID 18195237